CLINICAL TRIAL: NCT02591030
Title: Randomised Phase II/III Study, Assessing the Safety and Efficacy of Modified Folfirinox Versus Gemcis in Locally Advanced, Unresectable and/or Metastatic Bile Duct Tumours
Brief Title: Safety and Efficacy of Modified Folfirinox Versus Gemcis in Bile Duct Tumours
Acronym: AMEBICA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408212; 2015-002282-35 (EudraCT Number)
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Bile Duct Cancer
Keywords: Bile Duct Cancer; phase II/III; Modified folfirinox; Gemcis
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEMCIS (Placebo Comparator)
  Interventions: Drug: GEMCIS
- mFOLFIRINOX (Experimental)
  Interventions: Drug: mFolfirinox

INTERVENTIONS:
Drug: GEMCIS — At D1 and D8 of each cycle, i.e. every 21 days for 6 months:
  * Cisplatin 25 mg/m² over 1 hour at D1 and D8
  * Gemcitabine 1000 mg/m² over 30 minutes at D1 and D8.
  Arms: GEMCIS
Drug: mFolfirinox — At D1 of each cycle, i.e. every 15 days for 6 months:
  * Oxiplatin: 85 mg/m² (IP/120 minutes)
  * Irinotecan: 180 mg/m² (IV/90 minutes)
  * Folinic acid: 400 mg/m² (or 200 mg/m² if Elvorine [calcium levofolinate]) (IV/2 hours), via a Y connector at the same time as irinotecan
  * 5-FU: 2400 mg/m² (IV over 46 hours) without 5FU bolus at D1
  Arms: mFOLFIRINOX

SUMMARY:
Bile duct tumours are rare. They are the 6th most common type of digestive cancer. Their therapeutic management is complex and must be multidisciplinary in nature. Most of the time, an endoscopic or radiological biliary drainage is necessary before any tumour treatment.

Their prognosis is poor due to the fact that they are normally diagnosed late, which makes curative surgery impossible. A population study in the Côte d'Or region of France reported a survival rate at 5 years of approximately 10%.

For the locally advanced or metastatic forms, treatment has not been properly codified. With respect to chemotherapy, prospective studies, most often phase II, are difficult to interpret due to a limited number of patients and due to the heterogeneity of this type of tumour (bile duct and pancreas tumours). Treatment with 5FU alone provides an objective response in approximately 10% of cases. In combination with mitomycin or carboplatin, the objective response rate is 20%, with a median survival period of 5 months. Interferon combined with 5FU has a better response rate (30%), but occurrences of different types of toxicity are more frequent.

More recently, gemcitabine and the 5FU-cisplatin combinations demonstrated objective tumour control in 50% of patients with a median survival period of 10 months. Gemcitabine combined with oxiplatin or with cisplatin has shown the same response rate but a median survival period of approximately 12 months.

The benefit of this combination has been confirmed in a phase III trial that compared the gemcitabine-cisplatin combination to gemcitabine alone, in 410 patients with locally advanced unresectable and/or metastatic bile duct cancer. The results were in favour of the combined treatment with a median survival period of 11.7 months (versus 8.1 months - HR 0.64 [0.52 - 0.80]). This combination is currently the reference first-line treatment.

DETAILED DESCRIPTION:
At the same time as these results, triple therapies involving 5FU + oxiplatin + irinotecan have objectively shown a significant increase in overall survival of patients with metastatic pancreatic adenocarcinoma compared to gemcitabine alone (median of 11.1 months versus 6.8 months, HR = 0.57 [0.45 - 0.73] p < 0.0001). The response rate and progression-free survival (PFS) have also been improved with these triple therapies; the response rates were 31.6% versus 9.4% p < 0.001 and the median PFS 6.4 months versus 3.3 months p < 0.001, respectively.

The adverse events observed with the triple therapy occurred more frequently, for febrile neutropaenia (5.4%), with the need to treat with growth factors (G-CSF for 42.5% of patients). Haematological and digestive toxicity was also higher: grade 3-4 neutropaenia was observed for 45.7% of patients in the FOLFIRINOX arm and 18.7% of patients in the gemcitabine arm (p = 0.0001); vomiting was noted for 14.5% of patients in the FOLFIRINOX arm and 4.7% in the gemcitabine arm (p = 0.002). Quality of life was improved in the FOLFIRINOX arm.

Due to the histological, therapeutic and prognostic similarities between pancreatic and bile duct cancer, it is interesting to assess this triple therapy compared to the current reference treatment in bile duct cancers: gemcitabine combined with cisplatin (GEMCIS). Due to the known higher levels of toxicity for this triple therapy (digestive and haematological), the investigators modified the conventional FOLFIRINOX regimen (mFOLFIRINOX) by removing the 5-FU bolus at D1 of each cycle. This modification to the regimen would appear not to decrease the efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* - WHO 0 or 1
* Age ≥ 18 years
* Tumour of the intrahepatic or extrahepatic (and/or hilar) bile ducts, or of the gallbladder
* Measurable abdominal metastases (at least a lesion >10 mm) and/or measurable, unresectable primary tumour
* Disease proven by histopathology or cytology (on metastasis or primary tumour)
* If there are no abdominal metastases, the unresectability must be confirmed by a hepatobiliary surgeon in a multidisciplinary team (MDT) meeting
* Bilirubin <1.5 N (after endoscopic or trance hepatic optimum biliary drainage, if necessary), AST and ALT <10N
* Serum creatinine <130 µmol/L, creatinine clearance >60 mL/min
* Neutrophils ≥ 1500/mm3 and platelets ≥ 75,000/mm3
* Prothrombin index > 70%
* Serum albumin > 25 g/L
* Patient registered with a social security scheme (including CMU)
* Signed informed consent form

Exclusion Criteria:

* - Non-measurable metastases and primary tumour
* Ampullary carcinoma or cancer of the pancreas with infiltration of the bile ducts or mixed tumours (hepatocholangiocarcinoma)
* Chemotherapy and/or radiotherapy within the last 4 months
* Other malignant tumour except in situ basal cell carcinoma or curatively treated carcinoma of the uterine cervix or other malignant tumour that has been treated and has been considered cured for at least 5 years
* Major comorbidity factors (unstable angina, myocardial infarction that has occurred within the last 6 months, heart failure ≥2 according to the NYHA classification, uncontrolled high blood pressure)
* Woman who is pregnant or breastfeeding, or patient of either sex who is of childbearing age and not using an adequate contraceptive method
* Not able to undergo the trial medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
percentage of patients who are alive without radiological progession | up to 6 months
  In phase II, the primary endpoint is the percentage of patients alive without radiological progression (assessed according to the RECIST v1.1 criteria) at 6 months (after randomisation).
  Patients who are in radiological progression or who have died before the 6 months have elapsed will be considered a failure for the primary endpoint at 6 months (after randomisation).
  A medical review will be conducted to decide on patients without radiological progression at 6 months; in the light of their entire medical file, they may be considered a failure (i.e. in progression) or they may be considered to be truly non-assessable (a 5% surplus of patients has been planned for this situation).
overall survival | up to 6 years
  In phase III, the primary endpoint is overall survival. This is defined as the period between the date of randomisation and the date of death (regardless of the cause). Patients who are lost to follow-up will be censored at the end-point for the analysis, or at the date when they were last heard of.

SECONDARY OUTCOMES:
overall survival | up to 6 months
  In phase II, this is defined as the period between the date of randomisation and the date of death (regardless of the cause). Patients who are lost to follow-up will be censored at the end-point for the analysis, or at the date when they were last heard of.
Tumour response | up to 6 months
  In phase II, the best tumour response will be assessed across all the treatments and will be described using the figures for the different categories: complete response, partial response, stable, progression or non-assessable.
Tumour response | up to 6 years
  In phase III, the best tumour response will be assessed across all the treatments and will be described using the figures for the different categories: complete response, partial response, stable, progression or non-assessable.
Toxicity of the treatment assessed according to NCI-CTC v 4.0 | up to 6 months
  In phase II, different types of toxicity assessed according to NCI-CTC v 4.0. Type of toxicity : Haematological (platelets and Neutrophils), Non-haematological (except for nausea, vomiting and alopecia) and neurological (paraesthesia)
Toxicity of the treatment assessed according to NCI-CTC v 4.0 | up to 6 years
  In phase III, different types of toxicity assessed according to NCI-CTC v 4.0. Type of toxicity : Haematological (platelets and Neutrophils), Non-haematological (except for nausea, vomiting and alopecia) and neurological (paraesthesia)
Biliary complications | up to 6 years
  In phase III : angiocholitis, obstruction of the main bile ducts or biliary stent obstruction
Biliary complications | up to 6 months
  In phase II : angiocholitis, obstruction of the main bile ducts or biliary stent obstruction
quality of life (EORTC QLQ-C30 ) | up to 6 years
  EORTC QLQ-C30 quality of life. Quality-of-life assessments will be performed until progression of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Phelip, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (42):
- France (42):
  - Chu Picardie, Amiens
  - Ico Paul Papin, Angers
  - CH Victor Dupouy, Argenteuil
  - CH de la Côte Basque, Bayonne
  - CHRU Besançon, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint-André, Bordeaux
  - Polyclinique Nord, Bordeaux
  - Hôpital Duchenne, Boulogne-sur-Mer
  - Centre François Baclesse, Caen
  - Chu D'Estaing, Clermont-Ferrand
  - Hôpitaux Civils, Colmar
  - Ch Sud Francilien, Corbeil-Essonnes
  - Centre de radiothérapie et oncologie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - Hôpital Michallon, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Clinique du cap d'Or, La Seyne-sur-Mer
  - CH Le Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Centre Hospitalier de Longjumeau, Longjumeau
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Lyon Sud, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Centre Catherine de Sienne, Nantes
  - CHR Orléans, Orléans
  - HEGP, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint-Jean, Perpignan
  - CHU La Miletrie, Poitiers
  - CHU Reims, Reims
  - Centre Eugène Marquis, Rennes
  - Hôpital Drôme Nord, Romans-sur-Isère
  - Chu Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CH Saint-Jean de Luz, Saint-Jean-de-Luz
  - CH Saint-Quentin, Saint-Quentin
  - Ch Robert Morlevat, Semur-en-Auxois
  - CAC Paul Strauss, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phelip JM, Desrame J, Edeline J, Barbier E, Terrebonne E, Michel P, Perrier H, Dahan L, Bourgeois V, Akouz FK, Soularue E, Ly VL, Molin Y, Lecomte T, Ghiringhelli F, Coriat R, Louafi S, Neuzillet C, Manfredi S, Malka D; PRODIGE 38 AMEBICA Investigators/Collaborators. Modified FOLFIRINOX Versus CISGEM Chemotherapy for Patients With Advanced Biliary Tract Cancer (PRODIGE 38 AMEBICA): A Randomized Phase II Study. J Clin Oncol. 2022 Jan 20;40(3):262-271. doi: 10.1200/JCO.21.00679. Epub 2021 Oct 18. PMID 34662180